CLINICAL TRIAL: NCT02176395
Title: Multi-"Omics" Research of Danhong Injection to Treat Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DH20140604
Record Dates: First submitted 2014-06-20; First posted 2014-06-27 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Acute Stroke
Keywords: Acute Ischemic Stroke; Randomized Controlled Trial; Traditional Chinese Medicine; Proteomics
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — danhong; Honghua extract, Carthamus tinctorius

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Danhong injection (Experimental): Based on the standard medical care, 40ml of Danhong injection, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Drug: Danhong injection; Procedure: Standard medical care
- placebo (Placebo Comparator): Based on the standard medical care, 40ml of 0.9% saline as the placebo, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Procedure: Standard medical care; Drug: placebo
- healthy volunteer (No Intervention)

INTERVENTIONS:
Drug: Danhong injection — 40ml Danhong injection added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion
  Other Names: A kind of injection made from two kind of Chinese herbs: Salvia miltiorrhiza and Safflower.
  Arms: Danhong injection
Procedure: Standard medical care — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of acute ischemic stroke (2010), including medical care for vital signs, control of temperature, blood pressure and glucose, improving cerebral blood circulation, antiplatelet treatment and nutritional supportive care.
  Arms: Danhong injection; placebo
Drug: placebo — 0.9% saline added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion
  Arms: placebo

SUMMARY:
The purpose of this study is to explore the pharmacological mechanism of Danhong injection in the treatment of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male inpatients

   * Age: 18 - 70 years.
   * Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze, vision or neglect. Ischemic stroke is defined as an event characterized by the sudden onset of an acute focal neurologic deficit presumed to be due to cerebral ischemia after CT scan excludes hemorrhage.
   * Clinical diagnosis of "Xueyu Zheng" (Blood Stasis Syndrome) as the scores of Chinese medicine symptoms scales of "Xueyu Zheng" in ischemic stroke ≥ 20. The Chinese medicine symptoms scales of "Xueyu Zheng" is defined as following (1)hemiplegia-10,(2)numbness of limbs-10，(3) dark face-9,(4)purple or dark lip-8,(5)Roughness of skin-4, (6) pain with fixed point-5, (7) purple or dark tongue-10,(8)ecchymosis on tongue-10,(9)purple sublingual vessel-10,(10)varicose sublingual vessel-8,(11)unsmooth pulse-8,(12)intermittent pulse-1.
   * Onset of symptoms in 1 week prior to initiation of administration of study drug.
   * Clinical diagnosis of cerebral anterior circulation obstruction.
   * 4≤NIHSS<20.
   * Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relatives, or deferred where applicable, according to the regulatory and legal requirements of the participating centers.
2. Female or male healthy volunteer

   * Age: 18 - 70 years.
   * Medical history, physical examination, vital signs, electrocardiogram(ECG) and laboratory results (including renal function, hepatic function, et al)with no clinically significant findings.
   * Healthy volunteer is willing to participate voluntarily and to sign a written informed consent form. Informed consent will be obtained from each volunteer, according to the regulatory and legal requirements of the participating centers.

Exclusion Criteria:

1. Female or male inpatients

   * Evidence of intracranial hemorrhage (ICH) or other cerebral diseases (eg.vascular malformation, tumor, abscess or multiple sclerosis etc.)on the CT-or MRI-scan.
   * Patients with thrombolysis or endovascular treatment.
   * Known history of allergy or suspected allergic to the drug.
   * Blood glucose 2.8 or > 16.8 mmol / l under the treatment of diabetes or with severe complications due to diabetes (eg. peripheral neuropathy, diabetic gangrene).
   * Liver function impairment with the value of ALT or AST over 1.5-fold of normal value.
   * Renal dysfunction with the value of serum creatinine over 1.5-fold of normal value.
   * Severe cardiac dysfunction on echocardiogram or the grade of heart function over Ⅲ grade.
   * History of prior stroke with mRS ≥2.
   * Complicated with atrial fibrillation.
   * Severe stroke as assessed by appropriate imaging techniques (eg. massive cerebral infarction including more than one lobe of brain or over 1/3 of blood-supply area of middle cerebral artery).
   * Prior disable patients.
   * Hemorrhagic tendency or recent severe or dangerous bleeding in 3 months.
   * Suspected addicted into alcohol or drug abuse.
   * With severe complications that would make the condition more complicated assessed by the investigator.
   * Woman with pregnancy, lactation or positive result of pregnancy test, or women who want to be pregnant in recent 6 months.
   * Woman who is under menstrual period.
   * Patient who is participating in other trials or has been participated in other trials in recent 3 months.
2. Healthy volunteer

   * Had a known history of chronic diseases including stroke, heart diseases, diabetes, COPD, Neuropsychiatric diseases and chronic infectious diseases, etc.
   * Coagulation disorders.
   * Conditions with increased bleeding risk.
   * Trauma or surgery in the 6 months prior to the study.
   * Use of any medication 4 weeks prior to the trial.
   * History of drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale 0-1 (favourable outcome) at Day 90 | Day 90

OTHER OUTCOMES:
The changes of serum proteomics in 36 patients selected from certain center | Day 0, Day 14, Day 90
  We wish to identify protein biomarkers in the blood that changed with Danhong treatment
The microRNA profile in 10 healthy volunteer | Day0
The mRNA profiles in 10 healthy volunteer | Day0
The proteomics profiles of 10 healthy volunteer | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhong, Professor, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Zhao Xingquan, Professor, Principal Investigator — Beijing Tiantan Hospital; Wang Yongyan, Professor, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Jiang Zhilin, Professor, Principal Investigator — 202 Military Hospital of China
Locations (4):
- China (4):
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Panjin Central Hospital, Panjin, Liaoning
  - 202 Military Hospital of China, Shenyang, Liaoning
  - Affiliated Hospital of Chifeng University, Chifeng, Neimenggu